CLINICAL TRIAL: NCT01507194
Title: A Multicenter, Randomized, Single-blind, Active-controlled, Parallel Group, Phase II Study to Evaluate the Efficacy, Safety, and Tolerability of a Single Intravenous (6 mg, 12 mg, 18 mg, 24 mg or 36 mg) Dose of the Neurokinin-1 Receptor Antagonist, Vestipitant (GW597599), Compared With a Single 4 mg Intravenous Ondansetron Hydrochloride Dose for the Treatment of Breakthrough Post-Operative Nausea and Vomiting After Failed Prophylaxis With an Ondansetron-Containing Regimen in Patients Undergoing Non-Emergency Surgical Procedures
Brief Title: A Study of Vestipitant (GW597599) in the Treatment of Breakthrough Postoperative Nausea and Vomiting (PONV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Accenture (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VNK115640
Record Dates: First submitted 2012-01-04; First posted 2012-01-10 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron; vestipitant

STUDY DESIGN:
Who Masked: Investigator

ARMS (6):
- Ondansetron 4 mg (Active Comparator)
  Interventions: Drug: Ondansetron
- Vestipitant 6 mg (Experimental)
  Interventions: Drug: Vestipitant
- Vestipitant 12 mg (Experimental)
  Interventions: Drug: Vestipitant
- Vestipitant 18 mg (Experimental)
  Interventions: Drug: Vestipitant
- Vestipitant 24 mg (Experimental)
  Interventions: Drug: Vestipitant
- Vestipitant 36 mg (Experimental)
  Interventions: Drug: Vestipitant

INTERVENTIONS:
Drug: Ondansetron — Single IV dose
  Other Names: Zofran
  Arms: Ondansetron 4 mg
Drug: Vestipitant — Single IV dose
  Other Names: GW597599
  Arms: Vestipitant 12 mg; Vestipitant 18 mg; Vestipitant 24 mg; Vestipitant 36 mg; Vestipitant 6 mg

SUMMARY:
This study will evaluate single IV doses of Vestipitant (GW597599) compared to 4 mg IV ondansetron for treating breakthrough postoperative nausea and vomiting (PONV) after failure of PONV prophylaxis with a regimen that includes 4 mg IV ondansetron.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female post-operative surgical subjects between the ages of 18-75 years.
* Female subject is of non-childbearing potential or of child-bearing potential and agrees to use specified contraception methods.
* Has 3 or more of the following independent risk factors for PONV: female gender; non-smoker; history of PONV or motion sickness; or planned post- operative opioids.
* Has received one dose of ondansetron as part of a PONV prophylaxis regimen for the surgical procedure.
* Has received general anesthesia.
* Meets ASA Physical Status Classification of 1 or 2 without an "E" modifier preoperatively on the day of surgery and has hematology and blood chemistry values within acceptable limits for surgery.
* Is capable of giving written informed consent.
* Experiences breakthrough PONV defined as: post-operative nausea of ≥ 7 on the Nausea Numeric Rating Scale; nausea resulting in a subject request for an anti-emetic; or an episode of emesis or retching.

Exclusion Criteria:

* A history of HIV.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of Screening.
* An ALT or AST >2.5 x ULN at Screening.
* Pregnant or lactating females.
* The subject is scheduled to undergo a laparoscopic biopsy only.
* The subject has a history of or is scheduled to undergo cardiac/cardiothoracic surgery.
* The subject is scheduled to receive neuraxial anesthesia(e.g., epidural, spinal, or caudal anesthesia)or total IV anesthesia.
* The subject is scheduled to receive propofol for maintenance of anesthesia (propofol as an induction agent is allowed).
* The subject is scheduled to receive an NK1 inhibitor (aprepitant/fosaprepitant) as part of a PONV prophylaxis regimen for the surgical procedure.
* The subject is scheduled to have gastric contents suctioned continuously during the surgical procedure via a nasogastric tube, or a nasogastric or oral gastric tube during the post-operative period. A single pass at the beginning or at the end of the procedure, and intraoperative gastric suctioning of air, will be permitted.
* The subject received an investigational drug within 30 days or was scheduled to receive any investigational drug in addition to vestipitant during the study period.
* The subject has persistent or recurrent nausea and/or vomiting due to other etiologies, including, but not limited to, gastric outlet obstruction, hypercalcemia, active peptic ulcer, increased intracranial pressure, chemotherapy, or brain metastases.
* The subject received radiation therapy to the abdomen or the pelvis within 7 days prior to receiving study medications and/or received radiation therapy to the abdomen or the pelvis in the evaluation period.
* The subject has a history of wound dehiscence.
* The subject has a history of any other illness which might pose an unacceptable risk by administering study medication.
* The subject has any current or past medical condition (e.g., vagotomy) and/or required medication to treat a condition that could affect the evaluation of the study.
* The subject has a known contraindication or hypersensitivity to ondansetron or ondansetron injection, any scheduled anaesthetic or analgesic agents, vestipitant or any component of the vestipitant formulation including Captisol.
* The subject received medication with known or potential antiemetic activity after the induction of anaesthesia (during the intraoperative or post- operative period) other than the planned Study Treatment.
* Current or planned use of strong or moderate inhibitors of CYP3A within 7 days or inducers of CYP3A within 14 days prior to study medication administration.
* The subject is unwilling or unable to follow the procedures outlined in the protocol.
* The subject is mentally or legally incapacitated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Complete Response | 10 min. after infusion start through 24 hrs. or discharge
  No emesis and no further rescue medication

SECONDARY OUTCOMES:
Nausea Numeric Rating Scale (NNRS) | Pre-dose; 5, 10, 15 min. post-dose; q 15 min. through 2 hrs. post-dose; q 2 hrs. through 24 hrs. post-dose; and 5 days post-dose
No Emesis/Vomiting | Pre-dose; continuous through 24 hrs. post-dose; and 5 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Brigandi, MD, PhD, Study Director — GlaxoSmithKline
Locations (7):
- United States (7):
  - Helen Keller Hospital, Sheffield, Alabama
  - Precision Trials, Phoenix, Arizona
  - Visions Clinical Research, Boynton Beach, Florida
  - CAP Anesthesia (St. Elizabeth's Medical Center), Boston, Massachusetts
  - Wake Forest University Anesthesia at Forsyth Medical Center, Winston-Salem, North Carolina
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburg, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Kranke P, Thompson JP, Dalby PL, Eberhart LH, Novikova E, Johnson BM, Russ SF, Noble R, Brigandi RA. Comparison of vestipitant with ondansetron for the treatment of breakthrough postoperative nausea and vomiting after failed prophylaxis with ondansetron. Br J Anaesth. 2015 Mar;114(3):423-9. doi: 10.1093/bja/aeu376. Epub 2014 Dec 8. PMID 25488303